CLINICAL TRIAL: NCT05656079
Title: To Evaluate the Cardiac Safety of Pegylated Liposomal Doxorubicin Concurrently Plus Trastuzumab and Pertuzumab in the Adjuvant Setting for Early-stage HER-2-positive Breast Cancer: a Multicenter, Randomized Controlled Clinical Study
Acronym: easy laugh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pudong Hospital (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kazuma
Record Dates: First submitted 2022-12-11; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Epirubicin; Cyclophosphamide; Trastuzumab; pertuzumab; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pegylated liposomal doxorubicin；cyclophosphamide；trastuzumab；pertuzumab ；docetaxel (Experimental): Pegylated liposomal doxorubicin 35 mg/m2, i.v. d1 +Cyclophosphamide 600 mg/m2 , i.v. d1 +Trastuzumab (8 mg/kg loading dose at first day only, then 6 mg/kg), i.v. d1+Pertuzumab (840 mg loading dose at first day only, then 420 mg), i.v. d1 ； q3w, for 4 cycles followed by Docetaxel 75mg/m2 , i.v. d1+ Pertuzumab 420 mg, i.v. d1+Trastuzumab 6 mg/kg, i.v. d1； q3w, for 4 cycles.
  After the completion of adjuvant therapy, patients are required to receive a total of 1 year of treatment with trastuzumab combined with pertuzumab.
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Cyclophosphamid; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Docetaxel
- Epirubicin；cyclophosphamide f；docetaxel；trastuzumab；pertuzumab (Active Comparator): Epirubicin 90 mg/m2 , i.v. d1 +Cyclophosphamide 600 mg/m2 , i.v. d1； q3w, for 4 cycles followed by Docetaxel 75mg/m2 , i.v. d1+Trastuzumab (8 mg/kg loading dose at first day only, then 6 mg/kg), i.v. d1+Pertuzumab (840 mg loading dose at first day only, then 420 mg), i.v. d1； q3w, for 4 cycles.
  After the completion of adjuvant therapy, patients are required to receive a total of 1 year of treatment with trastuzumab combined with pertuzumab.
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamid; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin — Drug: Pegylated liposomal doxorubicin (35 mg/m2) will be administered by an intravenous infusion on day 1 of each21-day cycle.
  Other Names: duomeisu; Doxorubicin Hydrochloride Liposome Injection
  Arms: pegylated liposomal doxorubicin；cyclophosphamide；trastuzumab；pertuzumab ；docetaxel
Drug: Epirubicin — Drug: Epirubicin (90 mg/m2) will be administered by an intravenous infusion on day 1 of each 21-day cycle.
  Other Names: biaoroubixing
  Arms: Epirubicin；cyclophosphamide f；docetaxel；trastuzumab；pertuzumab
Drug: Cyclophosphamid — Drug: Cyclophosphamide (600 mg/m2) will be administered by an intravenous infusion on day 1 of each 21-day cycle.
  Other Names: huanlinxianan
Drug: Trastuzumab — Drug: Trastuzumab (8 mg/kg loading dose at first day only, then 6 mg/kg) will be administered by an intravenous infusion on day 1 of each 21-day cycle.
  Other Names: qutuozhudankang
Drug: Pertuzumab — Drug: Pertuzumab (840 mg loading dose at first day only, then 420 mg) will be administered by an intravenous infusion on day 1 of each 21-day cycle.
  Other Names: patuozhudankang
Drug: Docetaxel — Drug: Docetaxel (75mg/m2) will be administered by an intravenous infusion on day 1 of each 21-day cycle.
  Other Names: duoxitasai

SUMMARY:
To evaluate the safety and efficacy of pegylated liposomal doxorubicin/cyclophosphamide/trastuzumab/pertuzumab followed by docetaxel/ trastuzumab/pertuzumab compared with epirubicin/cyclophosphamide followed by docetaxel/trastuzumab/pertuzumab in the adjuvant treatment of early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old, Female;
2. Subjects with histopathologically confirmed invasive breast cancer;
3. HER2-positive breast cancer (Immunohistochemistry score of 3+ or fluorescence in situ hybridization positivity);
4. No distant metastasis;
5. Lymph node positive or negative, primary tumour≥2cm;
6. Lymph node negative，primary tumour≤2cm and any of the following factors; 1) Histological grade 3; 2) ER negative (<10%) and PR negative (<20%); 3) Age<35 years old; 4) Pathological hint: vascular invasion or intravascular cancer thrombus;
7. Surgery was completed and chemotherapy was started within 8 weeks after surgery;
8. Before and after chemotherapy LVEF≥55%;
9. ECOG performance status of 0-1;
10. Signed the informed consent.

Exclusion Criteria:

1. Subjects who are known to be allergic or intolerant to chemotherapy drugs or their excipients;
2. Previously suffered from invasive breast cancer, and other malignant tumors within 5 years (excluding carcinoma in situ of the cervix, carcinoma in situ of the rectum, carcinoma in situ of melanoma, basal cell carcinoma of the skin, and squamous cell carcinoma);
3. For breast cancer, have received any anti-tumor therapy before randomization (except surgical treatment before enrollment);
4. Hematopoietic function, renal function and liver function meet one of the following conditions: 1) Neutrophil count ≤1.5×109/L; 2) Platelet count ≤ 50×109/L; 3) Hemoglobin ≤ 8.0g/dL; 4) Creatinine clearance rate ≤30ml/min; 5) AST and ALT ≥ 2.5 times the upper limit of normal in subjects without liver metastases; 6) Bilirubin ≥ 2 times the upper limit of normal; 7) APTT/PT≥1.5 times the upper limit of normal;
5. Have a history of cardiovascular disease or associated with severe cardiovascular disease, lung disease;
6. Active hypertension: systolic blood pressure ≥ 180mmHg, diastolic blood pressure ≥ 90mmHg;
7. NYHA cardiac insufficiency grading ≥ Ⅲ grade;
8. Severe, uncontrollable systemic disease;
9. Subjects who are pregnant or breastfeeding, or subjects who cannot ensure effective contraceptive measures during the study treatment;
10. Subjects who participated in other clinical trials at the same time;
11. Subjects determined by the investigator to be inappropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
1-year incidence of cardiotoxicity | 1-year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pudong Hospital, Shanghai, China